CLINICAL TRIAL: NCT03196635
Title: Patient-Assisted Compression - Impact on Image Quality and Workflow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 124.03-2017-GES-0002
Record Dates: First submitted 2017-06-19; First posted 2017-06-23 (Actual); Results first posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- All Study Participants (Experimental): All subjects will undergo their regularly scheduled full-field digital mammogram, consisting of bilateral, 2-view (craniocaudal [CC] and mediolateral oblique [MLO]) image acquisition. In addition, a study-specific, unilateral 2-view image set will obtained, utilizing the PA breast compression mode.
  Interventions: Device: Patient-Assisted (PA) Breast Compression; Device: Technologist-Controlled (TC) Breast Compression

INTERVENTIONS:
Device: Patient-Assisted (PA) Breast Compression — The technologist will properly position the breast and apply minimum compression. The subject will be instructed to apply compression as the technologist ensures the breast tissue is in appropriate position and tautness. The technologist will then guide the subject to achieve appropriate compression level, sufficient but not excessive, and the image will be acquired. This will be done for both standard views CC & MLO.
Device: Technologist-Controlled (TC) Breast Compression — TC compression will be conducted per standard of care practices at the site.

SUMMARY:
This study is being conducted to compare the image quality of breast images obtained using standard (technologist-controlled [TC]) compression and patient-assisted (PA) compression and to evaluate the impact of PA compression on clinical workflow.

DETAILED DESCRIPTION:
Patient-assisted (PA) compression allows the patient to participate in controlling the amount of compression force during mammography and is a personalized approach that has demonstrated successful reduction in discomfort experienced during mammography. GE Healthcare's Senographe Pristina, an innovative mammography platform that provides both two-dimensional (2D) and three-dimensional (3D) imaging capabilities, offers both standard and PA compression modes. This study is being conducted to compare the image quality of breast images obtained using TC compression and PA compression, and to evaluate the impact of PA compression on clinical workflow. The study population will consist of adult asymptomatic women presenting for screening 2D mammography.

ELIGIBILITY:
Inclusion Criteria:

* Are women aged 40 years or older;
* Are asymptomatic and scheduled for FFDM screening mammography;
* Have left and right breasts;
* Have breast sizes compatible with the dimensions of a 24 x 31 cm image detector, without anatomical cut-off;
* Are documented as non-pregnant based on the investigator's medical judgment and in consideration of local clinical practice standards for evidence of non-pregnancy;
* Are able and willing to comply with study procedures; and
* Are able and willing to provide written informed consent to participate.

Exclusion Criteria:

* Have been previously included in this study or are participating in another study expected to interfere with study procedures or outcomes;
* Have undergone diagnostic or surgical intervention(s) or procedure(s) on either breast, including breast biopsy, lumpectomy, or reconstruction, within five (5) years (≤ 5 years) of the study exam date;
* Are currently undergoing radiotherapy or chemotherapy, or have a history of prior radiotherapy treatment on either breast;
* Are currently lactating; or
* Have breast implants.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Asymptomatic women, aged 40 years or older scheduled for FFDM screening mammography
Enrollment: 31 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Schilling, Principal Investigator — Boca Raton Regional Hospital
Locations (1):
- Boca Raton Regional Hospital Christine E. Lynn Women's Health and Wellness Institute, Boca Raton, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: All subjects will undergo their regularly scheduled full-field digital mammogram, consisting of bilateral, 2-view (craniocuadal [CC] and mediolateral oblique [MLO]) image acquisition. In addition, a study-specific, unilateral 2-view image set will obtained, utilizing the patient-assisted breast compression mode.
Period: Overall Study
Arm/Group | All Study Participants
Started | 31
Completed | 30
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Subject population consisted of adult women (>/= 40 years of age) clinically indicated for an FFDM exam.
Groups:
- All Study Participants: All subjects will undergo their regularly scheduled full-field digital mammogram, consisting of bilateral, 2-view (CC/MLO) image acquisition. In addition, a study-specific, unilateral 2-view image set will obtained, utilizing the patient-assisted breast compression mode.
  Patient-Assisted Breast Compression: The technologist will properly position the breast and apply minimum compression. The subject will be instructed to apply compression as the technologist ensures the breast tissue is in appropriate position and tautness. The technologist will then guide the subject to achieve appropriate compression level, sufficient but not excessive, and the image will be acquired. This will be done for both standard views CC/MLO.
Arm/Group | All Study Participants
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 1
Breast of Interest [Count of Participants; unit: Participants] — One breast per eligible subject was randomly assigned as her 'breast of interest' which underwent study-specific procedures and image evaluations. Randomization of breast of interest was performed so that approximately half the subjects were assigned to the first breast imaged and the other half was assigned to the second breast imaged. The laterality of the breast of interest depended on which breast (left or right) the technologist imaged first and second in standard practice.
  Participants
    First breast of interest | 16
    Second breast of interest | 14
    Withdrawn subject | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Acceptable Overall Clinical Image Quality for Patient-assisted (PA) and Technologist-controlled (TC) Image Sets
Description: One PA image set and one TC image set was acquired from each completed subject. The overall clinical image quality acceptability was collected and summarized on a per subject-basis using binary responses of either acceptable or unacceptable for unilateral, two-view PA and TC compression image sets. Two readers evaluated each of the 60 image sets (30 PA and 30 TC compression image sets from 30 completed participants). In cases of disagreement between Readers 1 and 2, a third reader provided adjudication.
Time Frame: Through study completion, on average 1 month
Population: 60 image sets (30 PA and 30 TC compression image sets from 30 participants) were evaluated for acceptability of overall clinical image quality by two readers. The one (1) withdrawn subject did not undergo image acquisition study procedures and thus was not included in this analysis set.
Measure: Count of Participants; unit: Participants
Groups:
- All Study Participants, PA Compression Image Sets: All image sets (30 patient-assisted compression image sets) were evaluated for acceptability of overall clinical image quality by two (2) readers.
- All Study Participants, TC Compression Image Sets: All image sets (30 TC compression image sets) were evaluated for acceptability of overall clinical image quality by two (2) readers.
Arm/Group | All Study Participants, PA Compression Image Sets | All Study Participants, TC Compression Image Sets
Number analyzed (Participants) | 30 | 30
Participants | 30 | 30

2. Secondary Outcome: Repeat Image Acquisition
Description: Number of incidences per image set when the technologists or readers indicated a repeat acquisition for PA and TC compression modes. More than one incident (i.e. reason for repeat from technologist or view indicated for repeat by readers) could have been selected for a given image set.
Time Frame: Through study completion, on average 1 month
Population: Instances of repeat imaging for each subject's PA (N=30) and TC (N=30) image sets were indicated by technologists during image acquisitions and by readers during image evaluations. The one withdrawn subject did not undergo image acquisition study procedures and thus was not included in this analysis set.
Measure: Count of Units; unit: Image sets
Units Other Than Participants: Image sets
Groups:
- All Study Participants, PA Compression Image Sets: Repeat imaging for PA compression image sets were indicated for each subject by technologists during image acquisitions and by readers during image evaluations.
- All Study Participants, TC Compression Image Sets: Repeat imaging for TC compression image sets were indicated for each subject by technologists during image acquisitions and by readers during image evaluations.
Arm/Group | All Study Participants, PA Compression Image Sets | All Study Participants, TC Compression Image Sets
Number analyzed (Participants) | 30 | 30
Number analyzed (Image sets) | 30 | 30
Image sets
  Technologist-indicated Repeat | 2 | 7
  Reader-indicated Repeat | 4 | 4

3. Secondary Outcome: Acceptability of Mammographic Attributes
Description: Acceptability of mammographic attributes using a binary response of either acceptable or unacceptable for unilateral, two-view PA and TC compression image sets were summarized.
Time Frame: Through study completion, on average 1 month
Population: The PA and TC image sets for all 30 subjects were evaluated for acceptability of pre-defined set of mammography attributes by Readers 1 and 2. Adjudication was not required if there was disagreement between the readers. The one withdrawn subject did not undergo image acquisition study procedures and thus was not included in this analysis set.
Measure: Number; unit: image sets
Groups:
- All Study Participants, PA Compression Image Sets: All image sets (30 PA compression image sets) were evaluated for acceptability of specific mammographic attributes by two (2) readers. Both readers evaluated all image sets from all available subjects.
- All Study Participants, TC Compression Image Sets: All image sets (30 TC compression image sets) were evaluated for acceptability of specific mammographic attributes by two (2) readers. Both readers evaluated all image sets from all available subjects.
Arm/Group | All Study Participants, PA Compression Image Sets | All Study Participants, TC Compression Image Sets
Number analyzed (Participants) | 30 | 30
image sets
  Acceptable Breast Positioning | 30 | 29
  Acceptable exposure and visualization of tissue | 30 | 30
  Acceptable breast compression | 30 | 30
  Acceptable image contrast | 30 | 30
  Acceptable sharpness of the image | 30 | 30
  Acceptable tissue visibility at the skin line | 30 | 30
  Acceptable noise level of the image | 30 | 30
  Acceptable artifacts level | 30 | 30

4. Other Pre Specified Outcome: Comparison of Image Acquisition Time
Description: The length of time it takes for image acquisition using each compression mode (TC Compression and PA Compression) were compared.
Time Frame: Through study completion, on average 1 month
Population: Imaging time was collected for each image set. 4 image sets were excluded from TC analysis due to repeat imaging per standard of care; repeat imaging wasn't allowed for PA compression. 1 subject's PA & TC image sets were excluded from analysis due to a protocol deviation. 1 withdrawn subject did not undergo imaging, so was not part of the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- All Study Participants, PA Compression Image Sets; All Study Participants, TC Compression Image Sets: Total image acquisition time was collected for each image set
Arm/Group | All Study Participants, PA Compression Image Sets | All Study Participants, TC Compression Image Sets
Number analyzed (Participants) | 29 | 25
minutes | 3.9 (1.0) | 3.4 (1.0)

5. Other Pre Specified Outcome: Technologist Interventions in PA Compression
Description: Data will be collected regarding any interventions made by the technologist during PA compression and this data were summarized.
Time Frame: Through study completion, on average 1 month
Population: Subjects underwent PA compression on their assigned Breast of Interest. Technologists were asked to provide confirmation if any intervention was necessary while the subject was controlling the compression. The one withdrawn subject did not undergo image acquisition study procedures and thus was not included in this analysis set.
Measure: Count of Participants; unit: Participants
Groups:
- All Study Participants: Technologists were asked to document if any intervention on compression was required during the PA compression procedures. If so, clarification regarding what type of intervention was performed was requested.
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
Participants
  Technologist had to increase compression | 0
  Technologist had to decrease compression | 1
  No intervention required | 29

6. Other Pre Specified Outcome: Compression Force for PA and TC Compressions
Description: Compression forces (decanewton [daN]) for each compression mode (TC and PA compression) were summarized for craniocaudal (CC) and mediolateral oblique (MLO) views. For each subject, both views were collected using both compression modes.
Time Frame: Through study completion, on average 1 month
Population: Compression force (daN) was captured for each view under each compression for all subjects. The one withdrawn subject did not undergo image acquisition study procedures and thus was not included in this analysis set.
Measure: Mean (Standard Deviation); unit: daN
Units Other Than Participants: Image Views
Groups:
- All Study Participants, PA Compression Image Sets: Compression force (daN) was captured for each view under Patient-Assisted Compression.
- All Study Participants, TC Compression Image Sets: Compression force (daN) was captured for each view under Technologist Compression.
Arm/Group | All Study Participants, PA Compression Image Sets | All Study Participants, TC Compression Image Sets
Number analyzed (Participants) | 30 | 30
Number analyzed (Image Views) | 60 | 60
daN
  CC | 9.1 (3.0) | 8.3 (2.0)
  MLO | 8.2 (2.7) | 8.7 (2.2)

7. Other Pre Specified Outcome: Breast Thickness for PA and TC Compressions
Description: Breast thickness (millimeter [mm]) for each compression mode (TC and PA compression) were summarized for craniocaudal (CC) and mediolateral oblique (MLO) views. For each subject, both views were collected using both compression modes.
Time Frame: Through study completion, on average 1 month
Population: Breast thickness (mm) was captured for each view under each compression for all subjects. The one withdrawn subject did not undergo image acquisition study procedures and thus was not included in this analysis set.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Image Views
Groups:
- All Study Participants, PA Compression Image Sets: Breast Thickness (mm) was captured for each view under PA Compression.
- All Study Participants, TC Compression Image Sets: Breast Thickness (mm) was captured for each view under TC compression.
Arm/Group | All Study Participants, PA Compression Image Sets | All Study Participants, TC Compression Image Sets
Number analyzed (Participants) | 30 | 30
Number analyzed (Image Views) | 60 | 60
mm
  CC | 52.0 (14.3) | 53.2 (14.0)
  MLO | 54.6 (16.1) | 53.7 (15.1)

8. Other Pre Specified Outcome: Radiation Dose for PA and TC Compressions
Description: Radiation dose (entrance skin air kerma [ESAK] in milligray [mGy]) for each compression mode (TC and PA compression) were summarized for craniocaudal (CC) and mediolateral oblique (MLO) views. For each subject, both views were collected using both compression modes.
Time Frame: Through study completion, on average 1 month
Population: ESAK was captured for each view under each compression for all subjects. The one withdrawn subject did not undergo image acquisition study procedures and thus was not included in this analysis set.
Measure: Mean (Standard Deviation); unit: mGy
Units Other Than Participants: Image Views
Groups:
- All Study Participants, PA Compression Image Sets: ESAK (mGy) was captured for each view under PA Compression.
- All Study Participants, TC Compression Image Sets: ESAK (mGy) was captured for each view under TC compression.
Arm/Group | All Study Participants, PA Compression Image Sets | All Study Participants, TC Compression Image Sets
Number analyzed (Participants) | 30 | 30
Number analyzed (Image Views) | 60 | 60
mGy
  CC | 4.5 (2.4) | 4.7 (2.4)
  MLO | 4.9 (2.6) | 4.8 (2.4)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for the duration of subject participation in the study, which was less than 1 month. Each subject was followed for Adverse Events from the time she entered the imaging suite for her exam until the time she exited the imaging suite after the exam.
Description: The definition of adverse events and/or serious adverse events aligns with the definitions provided by clinicaltrials.gov.
Groups:
- All Study Participants: Except for one subject who withdrew from the study prior to imaging procedures, all subjects underwent their regularly scheduled full-field digital mammogram, consisting of bilateral, 2-view (CC and MLO) image acquisition. In addition, a study-specific, unilateral 2-view image set was obtained, utilizing the patient-assisted breast compression mode.
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT03196635/Prot_SAP_000.pdf